CLINICAL TRIAL: NCT03532568
Title: Klotho and Fibroblast Growth Factor 23 in Chronic Kidney Disease-associated Pruritus and Their Response to Narrowband Ultraviolet B
Brief Title: Klotho in Chronic Kidney Disease-associated Pruritis (CKD-aP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, principal investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Dermatology 8
Record Dates: First submitted 2018-04-26; First posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Chronic Kidney Disease-associated Pruritus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CKD-aP patients (Experimental): skin biopsy for Klotho and fibroblast growth factor 23 levels in skin tissue and their response to narrow band ultraviolet B
  Interventions: Other: skin biopsy; Radiation: narrowband ultraviolet B
- CKD patients without pruritis (Experimental): skin biopsy for Klotho and fibroblast growth factor 23 levels in skin tissue
  Interventions: Other: skin biopsy
- normal healthy participants (Experimental): skin biopsy for Klotho and fibroblast growth factor 23 levels in skin tissue
  Interventions: Other: skin biopsy

INTERVENTIONS:
Other: skin biopsy — 4mm punch skin biopsy
Radiation: narrowband ultraviolet B — narrowband ultraviolet B for CKD-aP patients
  Arms: CKD-aP patients

SUMMARY:
Studying whether Klotho and FGF23 have a role in UP and whether their expression change by BB-UVB with the improvement of pruritus.

DETAILED DESCRIPTION:
Uremic pruritus (UP), also known as Chronic Kidney Disease-associated pruritus (CKD-aP), is the most common cause of Generalized Pruritus (GP). UP is multifactorial; not due to a single cause but as a result of combined action of multiple factors. UP has a major clinical impact because it is strongly associated with poor quality of life, impaired sleep, depression, and increased mortality. UP patient always feels he is drained and distressed.

Alpha Klotho is the protein product of the anti-aging klotho gene. This protein exists in two forms: soluble Klotho (s-Klotho) and membranous Klotho (m-Klotho). The kidney is the principal organ that produces, regulates, and metabolizes Klotho.

Membranous Klotho acts as a co-receptor to enhance the binding of fibroblast growth factor 23 (FGF23) to FGF receptors (FGFRs) through the formation of Klotho/FGFR/FGF23 complex. Interestingly, soluble Klotho can also bind to FGF23/FGFR, but it prevents high FGF23-induced toxicity.

In chronic kidney disease( CKD), soluble Klotho is still detectable although it is much lower than in healthy human beings, suggesting that it is produced from extrarenal organ(s) or tissue(s) not yet identified which may be the skin.

FGF23 is a peptide released from bone tissue osteocytes and osteoblasts. It plays an important role in the bone-kidney axis and the regulation of calcium and phosphate homeostasis. In CKD, Klotho is linearly decreased prior to the rise of FGF23 so it is considered a biomarker for early detection of kidney damage.

Klotho deficiency contributes to vascular and soft-tissue calcification in CKD patients. In CKD-aP patients, there is metastatic micro-calcification due to calcium deposition in skin and this is one of the etiological causes of UP. Whether Klotho has a role in this assumption is still unclear.

Phototherapy is a proven method for the management of many pruritic disorders. Narrowband ultraviolet B (NB-UVB) can be considered as a feasible treatment option for CKD-aP. One of its possible mechanisms is the reduction of skin calcium-ion content. Whether this is via changing Klotho expression is still unknown.

Therefore, our study aims at knowing whether Klotho and FGF23 have a role in UP and whether their expression change by NB-UVB with the improvement of pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD on dialysis.
* Age >18 years old.
* Both sexes.

Exclusion Criteria:

* Age <18 years old.
* Any contraindication to phototherapy (e.g, past skin cancer) for those with pruritus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Estimation of tissue levels of Klotho and FGF23 by ELISA in chronic kidney disease-associated pruritis and chronic kidney disease patients and comparing them with healthy control subjects. | 6 months
Estimation of tissue levels of Klotho and FGF23 BY ELISA after treatment with narrowband ultraviolet B in chronic kidney disease-associated patients. | 6 months